CLINICAL TRIAL: NCT04613752
Title: Evaluation and Follow up of Diaphragm Function in Acute Respiratory Distress Syndrome Patients With Veino-venous Extracorporeal Oxygenation Membrane
Brief Title: Diaphragm Dysfunction in ARDS Patients With V-V ECMO
Acronym: DD-ECMO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No more Covid patients in the service and number of patients included sufficient for stastistical analysis.
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP190988
Record Dates: First submitted 2020-10-15; First posted 2020-11-03 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-05

CONDITIONS: Respiratory Distress Syndrome
Keywords: ARDS; ECMO; diaphragm function
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): A single experimental group in which diaphragmatic function measurements and diaphragmatic ultrasound will be performed.
  Interventions: Device: diaphragmatic function measurements and diaphragmatic ultrasound

INTERVENTIONS:
Device: diaphragmatic function measurements and diaphragmatic ultrasound — A single experimental group in which diaphragmatic function measurements and diaphragmatic ultrasound will be performed.

SUMMARY:
Use of veno-venous extracorporeal oxygenation membrane is a therapeutic option for the management of the most severe patients with acute respiratory distress syndrome (ARDS).

Given the prolonged duration of this strategy, the question of its impact on the occurrence on diaphragm dysfunction has been raised. The present study endeavors to evaluate and follow up the prevalence, risk factors and prognosis of diaphragm dysfunction in patients with VV-ECMO.

DETAILED DESCRIPTION:
Use of veno-venous extracorporeal oxygenation membrane is a therapeutic option for the management of the most severe patients with acute respiratory distress syndrome (ARDS). It allows to provide a protective lung ventilation by reducing the level of airway pressures generated by the ventilator. The objective is to minimize the harmful effects of mechanical ventilation in the lungs and to provide adequate gases exchanges. This strategy requires a deep sedation to allow a perfect synchrony between the patient and the ventilator. Such a synchrony puts the respiratory muscles - in particular the diaphragm - completely at rest.

Given the prolonged duration of this strategy, the question of its impact on the occurrence on diaphragm dysfunction has been raised. Such a dysfunction has been associated with prolonged duration of mechanical ventilation and poor outcomes but its effect in patients with veno-venous extracorporeal oxygenation membrane has never been evaluated so far.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* ARDS according to the Berlin definition
* V-V ECMO
* patient or next of kin agrees to participate
* patient with health insurance

Exclusion Criteria:

* pregnancy
* Opposition to participate
* Contra indications to the phrenic nerves stimulation technique (pace maker, pneumothorax)"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Diaphragm function | until day 28
  as defined by the pressure generating capacity of the diaphragm < 11 cmH2O

SECONDARY OUTCOMES:
Duration of ECMO | until day 60
  from inclusion until ECMO removal
Duration of invasive mechanical ventilation | until day 60
  from inclusion until extubation

CONTACTS AND LOCATIONS:
Overall Officials: Martin Dres, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Pitié-Salpêtrière, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gautier M, Joussellin V, Ropers J, El Houari L, Demoule A, Similowski T, Combes A, Schmidt M, Dres M. Diaphragm function in patients with Covid-19-related acute respiratory distress syndrome on venovenous extracorporeal membrane oxygenation. Ann Intensive Care. 2023 Sep 26;13(1):92. doi: 10.1186/s13613-023-01179-w. PMID 37752337